CLINICAL TRIAL: NCT04328285
Title: Chemoprophylaxis of SARS-CoV-2 Infection (COVID-19) in Exposed Healthcare Workers : A Randomized Double-blind Placebo-controlled Clinical Trial
Brief Title: Chemoprophylaxis of SARS-CoV-2 Infection (COVID-19) in Exposed Healthcare Workers
Acronym: COVIDAXIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: French authority's decision
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20PH061; 2020-001188-96 (EudraCT Number)
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; nasopharyngeal swab; pneumonia; Hydroxychloroquine; Lopinavir/ritonavir; Healthcare Workers
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Hydroxychloroquine; lopinavir-ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: A randomized double-blind placebo-controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (HCQ) vs Placebo (Experimental): Group 1.1: HCQ 200 mg : 2 tablets on the evening at Day 1 and 2 tablets on the morning at Day 2 and 1 tablet once daily afterwards
  Group 1.2: Placebo of HCQ, 2 tablets on the evening at Day 1 and 2 tablets on the morning at Day 2 and 1 tablet once daily afterwards.
  Interventions: Drug: Hydroxychloroquine; Drug: Placebo of Hydroxychloroquine
- Lopinavir/ritonavir (LPV/r) vs Placebo (Experimental): Group 2.1: LPV/r 200/50 mg, 2 tablets twice daily
  Group 2.2: Placebo of LPV/r, 2 tablets twice daily
  Interventions: Drug: Lopinavir and ritonavir; Drug: Placebo of LPV/r Tablets

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine Oral Tablets
  Other Names: Plaquenil
  Arms: Hydroxychloroquine (HCQ) vs Placebo
Drug: Placebo of Hydroxychloroquine — Placebo of Hydroxychloroquine Oral Tablets Placebo manufactured to mimic Hydroxychloroquine tablets
  Arms: Hydroxychloroquine (HCQ) vs Placebo
Drug: Lopinavir and ritonavir — LPV/r Oral Tablets
  Other Names: Kaletra
  Arms: Lopinavir/ritonavir (LPV/r) vs Placebo
Drug: Placebo of LPV/r Tablets — Placebo of LPV/r Oral Tablets Placebo manufactured to mimic LPV/r tablets
  Arms: Lopinavir/ritonavir (LPV/r) vs Placebo

SUMMARY:
Since December 2019, the emergence of a new coronavirus named SARS-Cov-2 in the city of Wuhan in China has been responsible for a major epidemic of respiratory infections, including severe pneumonia. Within weeks, COVID-19 became a pandemic.

In the absence of specific antiviral treatment, a special attention should be given to prevention. Personal protection equipments may be insufficiently protective, including in healthcare workers, a significant proportion of whom (around 4%) having been infected in the outbreaks described in China and more recently in Italy. Infection in healthcare workers could result from the contact with COVID-19 people in community or with infected colleagues or patients.

As it will take at least a year before vaccines against SARS-CoV-2 becomes available, chemoprophylaxis is an option that should be considered in this setting where prevention of SARS-CoV-2 infection in Health Care Workers.

The COVIDAXIS trial evaluates a chemoprophylaxis of SARS-CoV-2 infection in Health Care Workers. This trial is divided into two distinct studies that could start independently each with its own randomization process: COVIDAXIS 1 will study Hydroxychloroquine (HCQ) versus placebo; COVIDAXIS 2 will study Lopinavir/ritonavir (LPV/r) versus placebo.

Upon randomization healthcare workers (HCWs) involved in the management of suspected or confirmed COVID-19 cases will be assigned to one of the following 2 treatment groups:

DETAILED DESCRIPTION:
The study COVIDAXIS 1(Hydroxychloroquine (HCQ) versus placebo) will be realized on 600 participants and will be implemented first in as many centers as possible.

Upon randomization, with 1:1 allocation ratio, healthcare workers involved in the management of suspected or confirmed COVID-19 cases will be assigned to one of the following 2 treatment groups:

* Group 1.1: HCQ 200 mg : 2 tablets on the evening at Day 1 and 2 tablets on the morning at Day 2 and 1 tablet once daily afterwards
* Group 1.2: Placebo of HCQ, 2 tablets on the evening at Day 1 and 2 tablets on the morning at Day 2 and 1 tablet once daily afterwards.

The COVIDAXIS 2 (Lopinavir/ritonavir (LPV/r) versus placebo will be realized on 600 participants and will be implemented in already participating and newer centers in a second step (when LPV/r becomes available).

Upon randomization, with 1:1 allocation ratio, healthcare workers involved in the management of suspected or confirmed COVID-19 cases will be assigned to one of the following 2 treatment groups:

* Group 2.1: LPV/r 200/50 mg : 2 tablets twice daily
* Group 2.2: Placebo of LPV/r, 2 tablets twice daily

Participants will receive the randomized treatment for 2 months and will be followed upon a 2.5 months period.

NB: there is no randomization procedure for participant inclusion in either COVIDAXIS 1 or COVIDAXIS 2

ELIGIBILITY:
Inclusion Criteria:

* Adult healthcare workers (HCWs) (for instance physicians, nurses, assistant nurses, dentists, physiotherapists, midwives, etc.)
* HCW involved at the time of enrolment in the care and the management of patients with confirmed or suspected SARS-CoV-2 infection in hospital settings, in outpatient care settings or in geriatric long-term care facilities. These HCWs have prolonged or repeated close contact to these patients.
* HCW tested negative for HIV
* HCW affiliated to the French health insurance system
* HCW women of childbearing age with an effective contraception (ethinylestradiol-containing contraceptive pills are not regarded as effective in the context of LPV/r treatment - COVIDAXIS 2)
* Willing to comply to study design and the follow-up
* Consent form signed

Exclusion Criteria:

For COVIDAXIS 1:

* HCW with positive SARS-CoV-2 RT-PCR of nasopharyngeal swab at the inclusion visit.
* HCW with past history of confirmed SARS-CoV-2 infection
* HCW with positive SARS-CoV-2 serology at the inclusion visit
* HCW with comorbidities such as hypothyroidism that need hormonal substitution, or retinopathy or with prior intermittent porphyria, or chronic renal failure (glomerular filtration rate < 30mL/min) or prior hepatic failure or psoriasis.
* HCW with prior diagnosis of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* HCW with known hypersensitivity/allergy to HCQ
* HCW with baseline QTc interval > 450ms in men or > 460ms in women and QTc <320 ms (both gender)
* HCW with personal or family history of long QT syndrome, torsades de pointes, or sudden death
* Pregnant HCW
* Breastfeeding HCW
* HCW taking comedications known to have interactions with HCQ according to the official characteristics of the product

For COVIDAXIS 2:

* HCW with positive SARS-CoV-2 RT-PCR of nasopharyngeal swab at the inclusion visit.
* HCW with past history of confirmed SARS-CoV-2 infection
* HCW with positive SARS-CoV-2 serology at the inclusion visit
* HCW with comorbidities such as chronic HCV infection treated by direct antiviral drugs or with hypothyroidism that need hormonal substitution, or known to have hypercholesterolemia hypertriglyceridemiaor chronic renal failure (glomerular filtration rate < 30mL/min) or prior hepatic failure
* HCW with known hypersensitivity/allergy to LPV/r
* HCW with baseline QTc interval > 450ms in men or > 460ms in women and QTc <320 ms (both gender)
* HCW with personal or family history of long QT syndrome, torsades de pointes, or sudden death
* Pregnant HCW
* Breastfeeding HCW
* HCW taking comedications known to have interactions with LPV/r according to the official characteristics of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of an symptomatic or asymptomatic SARS-CoV-2 infection among healthcare workers (HCWs) | Up to 2.5 months
  An infection by SARS-CoV-2 is defined by either:
  * a positive specific Reverse Transcription - Polymerase Chain Reaction (RT-PCR) on periodic systematic nasopharyngeal swab during follow-up OR
  * a positive specific RT-PCR on a respiratory sample in case of onset of symptoms consistent with COVID-19 during follow-up OR
  * a seroconversion to SARS-CoV-2 after randomization.

SECONDARY OUTCOMES:
Evaluation of the occurrence of adverse events in each arm, | Up to 2.5 months
  Number of adverse events expected or unexpected, related and unrelated to the treatment, notably grades 2, 3 and 4 (moderate, severe and lifethreatening, according to the Adverse National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0) in each arm.
Evaluation of the discontinuation rates of the investigational drug in each arm, | Up to 2 months
  Number of treatment discontinuations in each arm
Evaluation of the adherence of participants to study drug, | Up to 2 months
  Treatment adherence rate will be assessed by:
  * measurement of LPV and HCQ plasma concentrations using LC-MS/MS or LC-Fluorimetric detection
  * the count of returned drugs at each visit.
Evaluation of the incidence of symptomatic cases of SARS-CoV-2 infection in each arm, | Up to 2.5 months
  Number of incident cases of symptomatic SARS-CoV-2 infections among HCWs in each arm.
  Symptomatic infection is defined as :
  * a positive specific RT-PCR on a respiratory or non respiratory sample OR
  * a thoracic CT scan with imaging abnormalities consistent with COVID-19.
  These investigations being performed in case of signs/symptoms consistent with COVID-19 during follow-up.
Evaluation of the incidence of asymptomatic cases of SARS-CoV-2 infection in each arm | Up to 2.5 months
  Number of incident cases of asymptomatic SARS-CoV-2 infection among HCWs in each randomization arm.
  Asymptomatic infection is defined as :
  * a positive specific RT-PCR on periodic systematic nasopharyngeal swab during clinical follow-up without consistent clinical signs/symptoms during follow-up OR
  * as seroconversion to SARS-CoV-2 between start and end of the study in HCWs that did not reported any consistent clinical symptoms during follow-up
Evaluation of the incidence of severe cases of SARS-CoV-2 infection in each arm. | Up to 2.5 months
  Number of incident cases of severe SARS-CoV-2 infections among HCWs in each randomization arm, defined as :
  * a positive specific RT-PCR on a respiratory sample OR
  * a thoracic CT scan with imaging abnormalities consistent with COVID-19 performed in case of onset of symptoms consistent with COVID-19 during follow-up in a participant who need to be hospitalized for respiratory distress. Respiratory distress defined as dyspnea with a respiratory frequency > 30/min, blood oxygen saturation <93%, partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300 and/or lung infiltrates >50% (1).
corrected QT interval (ms) | At baseline, at D2 (only for COVIDAXIS 1) and every week up to 2 months.
  Safety. Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Botelho-Nevers, MD, PhD, Principal Investigator — CHU de Saint-Etienne; Bruno Hoen, MD, PhD, Study Director — Institut Pasteur
Locations (9):
- France (9):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No